CLINICAL TRIAL: NCT02796378
Title: Living With Statins - The Impact of Cholesterol Lowering Drugs on Health, Lifestyle and Well-being
Brief Title: Living With Statins - Interventional Exercise Study
Acronym: LIFESTAT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Flemming Dela, Professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: LIFESTAT - Exercise study
Record Dates: First submitted 2016-05-27; First posted 2016-06-10 (Estimated); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Cardiovascular Disease; Diabetes Mellitus
Keywords: physical activity; statin therapy; diabetes mellitus; cardiovascular disease; Q10-supplementation
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Training+Simvastatin+Q10-placebo (Active Comparator): Training+Simvastatin+Q10-placebo. 8 Weeks of exercise training on a bicycle ergometer three times a week and 40 mg of Simvastatin pr day and Q10-placebo.
  Interventions: Drug: Training+Simvastatin+Q10-placebo
- Training+Simvastatin-placebo+Q10-placebo (Placebo Comparator): Training+Simvastatin-placebo+Q10-placebo. 8 Weeks of exercise training on a bicycle ergometer three times a week, Simvastatin-placebo and Q10-placebo.
  Interventions: Drug: Training+Simvastatin-placebo+Q10-placebo
- Training+Simvastatin+Q10 (Active Comparator): Training+Simvastatin+Q10. 8 Weeks of exercise training on a bicycle ergometer three times a week and 40 mg of Simvastatin pr day in combination with 400 mg of oral supplementation with Q10.
  Interventions: Drug: Training+Simvastatin+Q10

INTERVENTIONS:
Drug: Training+Simvastatin+Q10-placebo — 8 weeks of exercise training on a bycycle ergometer 3 times/week combined with Simvastatin 40 mg/day and Q10-placebo.
  Other Names: SP
  Arms: Training+Simvastatin+Q10-placebo
Drug: Training+Simvastatin-placebo+Q10-placebo — 8 weeks of exercise training on a bycycle ergometer 3 times/week combined with Simvastatin-placebo and Q10-placebo.
  Other Names: PL
  Arms: Training+Simvastatin-placebo+Q10-placebo
Drug: Training+Simvastatin+Q10 — 8 weeks of exercise training on a bycycle ergometer 3 times/week combined with Simvastatin 40 mg/day and Q10 400 mg/day.
  Other Names: Simvastatin KRKA; SQ
  Arms: Training+Simvastatin+Q10

SUMMARY:
Background. Statins are cholesterol lowering drugs that are prescribed to lower the risk of cardio-vascular diseases. The use of statins has increased markedly and it is now one of the most prescribed drugs in the world. More than 600,000 people in Denmark are taking statins on a daily basis, approximately 40 % of these are taking the medication without having any other risk factors for cardio-vascular diseases than elevated blood-cholesterol i.e. they are in primary prevention.

Statins are not without side effects and studies have shown that there is an elevated risk of developing diabetes when taking statins. This has led to an increased debate about the use of statins in primary prevention. Furthermore a large meta-analysis has shown that to prevent one event of cardio-vascular disease, it is necessary to treat 200 people for 3-5 years. These data suggest that more conservative use of statins to prevent CVD in otherwise healthy individuals at low risk for future CVD may be warranted.

Other side effects of statins are muscle myalgia, muscle cramps and fatigue which potentially can prevent a physically active lifestyle. The biomedical background of these side effects is not fully elucidated but it has been shown that there is a link to decreasing levels of an important enzyme, Q10, which plays a role in muscle energy metabolism.

Hypothesis

The overarching research question is: why does statin treatment cause muscle pain? Does statin treatment impair (or even prohibit) physical exercise training? Furthermore the following questions will be investigated:

A. Does statin treatment cause:

1. Decreased muscle strength?
2. Skeletal muscle inflammation?
3. Decreased mitochondrial respiratory function? B. Abnormal glucose homeostasis?

Re question A & B: If so, can physical training counteract this effect of statin treatment?

DETAILED DESCRIPTION:
Background:

Hypercholesterolemia and statin use in Denmark

Simvastatin is the most commonly prescribed statin, a class of drugs that inhibit hydroxyl-methyl-glutaryl (HMG) coenzyme A reductase, and thereby blocking biosynthesis of cholesterol in the liver. Simvastatin is prescribed for individuals with elevated low-density lipoprotein cholesterol (LDL-C) and/or total cholesterol, because these clinical parameters are viewed as a risk factor for cardiovascular-disease (CVD), even in the absence of other health problems or risk factors, such as previous myocardial infarction, diabetes or hypertension.

Approximately 40% of the prescriptions for statins are issued for primary prevention of elevated cholesterol by general practitioners to patients without bodily symptoms or signs. Only the "cholesterol number" makes the risk of heart attack and stroke visible. The lack of symptoms is likely to be of importance for patients' adherence to treatment as is adverse effects. A number of factors, such as information in mass media and changes in daily life, may affect the decision to take the treatment

Treatment guidelines for hypercholesterolemia:

The guidelines indicate preventive treatment with statins is appropriate in individuals with >10% predicted risk of a major vascular event within 5 years, while, some, but not all opinion-leaders advocate a 5% threshold. Nevertheless, statin therapy failed to reduce all-cause mortality in a meta-study of 65,229 patients without CVD, some of whom had diabetes. Similarly, a Cochrane review analysis, which included some studies in which more than 10% of the patients had history of CVD, showed only 0.5% reduction in all-cause mortality, indicating that for every 200 patients taking statins daily for 5 years, 1 death would be prevented. These data suggest that more conservative use of statins to prevent CVD in otherwise healthy individuals at low risk for future CVD may be warranted.

The downside:

Rhabdomyolysis (skeletal muscle cell death) is an infrequent but serious side-effect of statin use, that can on rare occasion lead to acute renal failure and death (i.e., 1.5 deaths per 106 prescriptions). Statin use is much more frequently associated with muscle dysfunction, including myalgia (muscle pain), cramps, and weakness. The reported incidence of myalgia varies from 1% (pharmaceutical company reports) to as high as 75% in statin-treated athletes. Mild to severe myalgia is a strong disincentive to regular exercise, and because regular exercise is one of the critical life-style approaches to preventing CVD and reducing blood cholesterol, this is a significant down-side of statin use. Regular exercise is also effective in preventing and treating obesity and type 2 diabetes, which themselves are risk factors for CVD.

The mechanism behind the myalgia is not known. However, the investigators behind this study has recently demonstrated that muscle mitochondrial function is impaired with statin treatment and the Q10 protein may play a key role in this. In addition, the statins also negatively affect the glucose tolerance, increasing the risk of type 2 diabetes.

Research questions:

The overarching research question is: why does statin treatment cause muscle pain? Does statin treatment impair (or even prohibit) physical exercise training? Furthermore the following questions will be investigated:

A. Does statin treatment cause:

1. Decreased muscle strength?
2. Skeletal muscle inflammation?
3. Decreased mitochondrial respiratory function? B. Abnormal glucose homeostasis?

Re question A & B: If so, can physical training counteract this effect of statin treatment?

Methodology:

Cohort

Patients that fulfil defined inclusion and exclusion criteria will be recruited from General Practice clinics in Copenhagen and news paper advertisements. The vast majority of these patients are being assessed on basis of the HeartScore risk estimation system that offers direct estimation of the ten-year risk of fatal cardiovascular disease in a format suited to the constraints of clinical practice. A staggered recruitment will be implemented.

30 men (age: 40-70 years; BMI: 25-35 kg/m2) before initiation of a statin treatment as primary prevention are recruited. No other risk factors for CVD except elevated total cholesterol (>6 mmol/l) and/or elevated LDL cholesterol (>3,5 mmol/l) and mild hypertension (<160/100 mm Hg) must be present.

The patients will be allocated (randomization by drawing a lot) to one of three groups:

* Physical exercise training and Simvastatin 40 mg/day and Q10 placebo
* Physical exercise training and Simvastatin 40 mg/day and Q10 400 mg/day supplementation
* Physical exercise training, Simvastatin placebo and Q10 placebo

The intervention period is 8 weeks with a series of experimental days before and after.

Experimental days (identical before and after the interventions):

Information day: health examination, ECG and Maximal oxygen uptake take (VO2 max).

Day 1 (overnight fasting, approximately 5 hours):

* Dual energy x-ray absorptiometry (DXA) scan (body composition and body fat).
* Oral glucose tolerance test + score questionnaire for muscle pain/discomfort (incl. Visual Analog Scale)
* Isokinetic strength and Rate of Force Development (PowerRig and KinCom dynamometer).
* Repeated VO2-max-test

Day 2 (overnight fasting approximately 7 hours):

* Muscle biopsy, vastus lateralis
* 2 step Euglycemic, hyperinsulinaemic clamp.

Training programme All training is supervised and takes place at the department. The training is aerobic, bicycle ergometer training (45 min/session at 60-70% of VO2max) three times a week for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Elevated blood-cholesterol

Exclusion Criteria:

* Cholesterol-lowering drugs
* Diabetes Mellitus
* Cardiovascular disease such as arrythmia, ischaemic heart disease.
* Musculoskeletal disorders preventing the subject to perform physical training
* Mental disorders preventing the subject to understand the project description.

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-06; Primary Completion 2021-07 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Physical performance measured by VO2-max | 8 weeks
  Difference in physical performance measured by VO2-max (mlO2/min/kgBW) in the three different intervention groups.

SECONDARY OUTCOMES:
Myalgia measured by VAS | 8 weeks
  Difference in potential myalgia, measured by visual analog scale (VAS) between the three different intervention groups.
Difference in muscle strength measured by KinCom dynamometer and PowerRig | 8 weeks
  Difference in muscle strength between the three different intervention groups.
Difference in glucose metabolism measured by hyperinsulinemic euglycemic clamp | 8 weeks
  Difference in glucose metabolism between the three different intervention groups.
Difference in mitochondrial function measured by respirometry | 8 weeks
  Difference in mitochondrial function between the three different intervention groups.

CONTACTS AND LOCATIONS:
Overall Officials: Flemming Dela, MD, MDSci, Principal Investigator — University of Copenhagen
Locations (1):
- University of Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boushel R, Gnaiger E, Schjerling P, Skovbro M, Kraunsoe R, Dela F. Patients with type 2 diabetes have normal mitochondrial function in skeletal muscle. Diabetologia. 2007 Apr;50(4):790-6. doi: 10.1007/s00125-007-0594-3. Epub 2007 Feb 15. PMID 17334651
- [Background] Ebrahim S, Casas JP. Statins for all by the age of 50 years? Lancet. 2012 Aug 11;380(9841):545-7. doi: 10.1016/S0140-6736(12)60694-1. Epub 2012 May 17. No abstract available. PMID 22607823
- [Background] Larsen S, Hey-Mogensen M, Rabol R, Stride N, Helge JW, Dela F. The influence of age and aerobic fitness: effects on mitochondrial respiration in skeletal muscle. Acta Physiol (Oxf). 2012 Jul;205(3):423-32. doi: 10.1111/j.1748-1716.2012.02408.x. Epub 2012 Feb 11. PMID 22212519
- [Background] Larsen S, Nielsen J, Hansen CN, Nielsen LB, Wibrand F, Stride N, Schroder HD, Boushel R, Helge JW, Dela F, Hey-Mogensen M. Biomarkers of mitochondrial content in skeletal muscle of healthy young human subjects. J Physiol. 2012 Jul 15;590(14):3349-60. doi: 10.1113/jphysiol.2012.230185. Epub 2012 May 14. PMID 22586215
- [Background] Larsen S, Stride N, Hey-Mogensen M, Hansen CN, Andersen JL, Madsbad S, Worm D, Helge JW, Dela F. Increased mitochondrial substrate sensitivity in skeletal muscle of patients with type 2 diabetes. Diabetologia. 2011 Jun;54(6):1427-36. doi: 10.1007/s00125-011-2098-4. Epub 2011 Mar 18. PMID 21424396
- [Background] Larsen S, Stride N, Hey-Mogensen M, Hansen CN, Bang LE, Bundgaard H, Nielsen LB, Helge JW, Dela F. Simvastatin effects on skeletal muscle: relation to decreased mitochondrial function and glucose intolerance. J Am Coll Cardiol. 2013 Jan 8;61(1):44-53. doi: 10.1016/j.jacc.2012.09.036. PMID 23287371
- [Background] Singh P, Kohr D, Kaps M, Blaes F. Skeletal muscle cell MHC I expression: implications for statin-induced myopathy. Muscle Nerve. 2010 Feb;41(2):179-84. doi: 10.1002/mus.21479. PMID 19813190
- [Background] Cholesterol Treatment Trialists' (CTT) Collaborators; Mihaylova B, Emberson J, Blackwell L, Keech A, Simes J, Barnes EH, Voysey M, Gray A, Collins R, Baigent C. The effects of lowering LDL cholesterol with statin therapy in people at low risk of vascular disease: meta-analysis of individual data from 27 randomised trials. Lancet. 2012 Aug 11;380(9841):581-90. doi: 10.1016/S0140-6736(12)60367-5. Epub 2012 May 17. PMID 22607822
- [Background] Parker BA, Thompson PD. Effect of statins on skeletal muscle: exercise, myopathy, and muscle outcomes. Exerc Sport Sci Rev. 2012 Oct;40(4):188-94. doi: 10.1097/JES.0b013e31826c169e. PMID 23000957
- [Background] Perk J, De Backer G, Gohlke H, Graham I, Reiner Z, Verschuren WM, Albus C, Benlian P, Boysen G, Cifkova R, Deaton C, Ebrahim S, Fisher M, Germano G, Hobbs R, Hoes A, Karadeniz S, Mezzani A, Prescott E, Ryden L, Scherer M, Syvanne M, Scholte Op Reimer WJ, Vrints C, Wood D, Zamorano JL, Zannad F; Comitato per Linee Guida Pratiche (CPG) dell'ESC. [European Guidelines on Cardiovascular Disease Prevention in Clinical Practice (version 2012). The Fifth Joint Task Force of the European Society of Cardiology and other societies on cardiovascular disease prevention in clinical practice (constituted by representatives of nine societies and by invited experts)]. G Ital Cardiol (Rome). 2013 May;14(5):328-92. doi: 10.1714/1264.13964. No abstract available. Italian. PMID 23612326
- [Background] Ray KK, Seshasai SR, Erqou S, Sever P, Jukema JW, Ford I, Sattar N. Statins and all-cause mortality in high-risk primary prevention: a meta-analysis of 11 randomized controlled trials involving 65,229 participants. Arch Intern Med. 2010 Jun 28;170(12):1024-31. doi: 10.1001/archinternmed.2010.182. PMID 20585067
- [Background] Ridker PM, Pradhan A, MacFadyen JG, Libby P, Glynn RJ. Cardiovascular benefits and diabetes risks of statin therapy in primary prevention: an analysis from the JUPITER trial. Lancet. 2012 Aug 11;380(9841):565-71. doi: 10.1016/S0140-6736(12)61190-8. PMID 22883507
- [Background] Taylor F, Ward K, Moore TH, Burke M, Davey Smith G, Casas JP, Ebrahim S. Statins for the primary prevention of cardiovascular disease. Cochrane Database Syst Rev. 2011 Jan 19;(1):CD004816. doi: 10.1002/14651858.CD004816.pub4. PMID 21249663